CLINICAL TRIAL: NCT00729677
Title: Prevalence of Delayed Nausea and Vomiting in Patients Being Treated With Oxaliplatin-based Regimens (mFOLFOX6 or FOLFOX7) for Colorectal Cancer
Brief Title: Delayed Nausea and Vomiting in Patients With Colorectal Cancer Receiving Oxaliplatin
Status: Completed | Type: Observational
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 237-04; BIMCP-NV-SURVEY; BIMCP-IRB-37-04; MERCK-BIMCP-NV-SURVEY
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Results first posted 2011-03-18 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer; Nausea; Vomiting
Keywords: nausea and vomiting; colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Nausea; Vomiting; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Learning how often patients experience nausea and vomiting after receiving anti-vomiting medicine and chemotherapy for colorectal cancer may help doctors plan better treatment and improve patients' quality of life.

PURPOSE: This clinical trial is studying delayed nausea and vomiting in patients with colorectal cancer receiving standard anti-vomiting medicine during the first course of chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the prevalence of delayed nausea and vomiting in patients with colorectal cancer receiving standard anti-emetic medications during the first course of an oxaliplatin-based chemotherapy regimen (mFOLFOX6 or FOLFOX7).

OUTLINE: This is a multicenter study.

Patients undergo collection of demographic, diagnostic, and treatment data at baseline. Patients complete the Functional Living Index-Emesis (FLIE) questionnaire at baseline prior to first chemotherapy infusion and at 5-7 days. Patients also fill out daily patient diaries about symptoms of nausea and vomiting, and use of medications to prevent these symptoms over days 1-5.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer
* Currently receiving OR scheduled to receive the first course of either of the following chemotherapy regimens:

  * mFOLFOX6
  * FOLFOX7
* No clinical or imaging evidence of brain metastasis

PATIENT CHARACTERISTICS:

* Able to maintain a diary and complete a standardized quality of life questionnaire in English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 90 days since prior aprepitant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiveing chemotherapy including oxaliplatin at the ambulatory care center
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2005-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Barry Fleishman, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center - Philipps Ambulatory Care Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original intent had been to analyze data on 100 chemotherapy cycles in 100 subjects. Instead, in order to accelerate accrual, we analyzed data on 1 cycle in 24 subjects and 2 cycles in 40 subjects.
Groups:
- Patients With Colorectal Cancer Starting Chemotherapy: patients starting chemotherapy for stage 3 or 4 colorectal cancer on regimens containing oxaliplatin. The chemotherapy is not part of the study but instead is initiated as standard care.
Period: Overall Study
Arm/Group | Patients With Colorectal Cancer Starting Chemotherapy
Started | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Colorectal Cancer Starting Chemotherapy
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Participants by Gender Who Reported Nausea During the First Week of Chemotherapy
Time Frame: Week 1 of FOLFOX chemotherapy
Measure: Number; unit: percentage of participants
Groups:
- Females: females starting chemotherapy for stage 3 or 4 colorectal cancer with regimens containing oxaliplatin. The chemotherapy is not part of the study but instead is initiated as standard care.
- Males: males starting chemotherapy for stage 3 or 4 colorectal cancer containing oxaliplatin. The chemotherapy is not part of the study but instead is initiated as standard care.
- Transgender: transgender subject starting chemotherapy for stage 3 or 4 colorectal cancer containing oxaliplatin. The chemotherapy is not part of the study but instead is initiated as standard care.
Arm/Group | Females | Males | Transgender
Number analyzed (Participants) | 28 | 35 | 1
percentage of participants | 64 | 34 | 100
Statistical Analysis 1: Comparison: Females vs Males vs Transgender; Test type: Superiority or Other; p = .05, ANOVA

2. Primary Outcome: Impact of Nausea and Vomiting on the Patient's Quality of Life as Measured by the Functional Living Index - Emesis Scale at 5-7 Days
Description: Scale describing impact of nausea and vomiting on quality of life on a seven-point Likert Scale with higher score indicating worse quality of life.
Time Frame: Week 1
Population: this data was not collected
Arm/Group | Patients With Colorectal Cancer Starting Chemotherapy
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants by History of Nausea Who Reported Nausea During the First Week of Chemotherapy
Description: Number of participants with factors associated with increased frequency of nausea in the first cycle of chemotherapy, including history of motion sickness, history of pregnancy-related morning sickness, history of prior chemotherapy, and history of nausea associated with prior chemotherapy
Time Frame: week 1
Measure: Number; unit: participants
Groups:
- Participants With History of Nausea: patients starting chemotherapy for stage 3 or 4 colorectal cancer receiving regimens containing oxaliplatin who had history of nausea.
- Participants With No History of Nausea: patients starting chemotherapy for stage 3 or 4 colorectal cancer receiving regimens containing oxaliplatin who had no history of nausea.
Arm/Group | Participants With History of Nausea | Participants With No History of Nausea
Number analyzed (Participants) | 23 | 41
participants
  nausea | 14 | 17
  No nausea | 9 | 24

4. Post Hoc Outcome: Number of Participants by Antiemetic Regimen Who Reported Nausea During First Cycle of Chemotherapy
Description: Number of participants on 2-drug (5HT3 inhibitor plus steroid) versus 3 drug (2-drug regimen plus an NK-1 inhibitor) who reported nausea during the first cycle of chemotherapy. 5HT-3 inhibitors included ondansetron, dolasetron, granisetron, and palonosetron. The NK-1 inhibitor was aprepitant. The steroid was dexamethasone.
Time Frame: Week 1
Measure: Number; unit: participants
Groups:
- Participants on 2-drug Regimen; Participants on 3-drug Regimen: patients starting chemotherapy for stage 3 or 4 colorectal cancer receiving 2-drug antiemetic regimens who reported nausea.
Arm/Group | Participants on 2-drug Regimen | Participants on 3-drug Regimen
Number analyzed (Participants) | 50 | 14
participants
  Reported nausea | 24 | 6
  No nausea | 26 | 8

ADVERSE EVENTS:
Arm/Group | Patients With Colorectal Cancer Starting Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 0/64

LIMITATIONS AND CAVEATS:
This was a convenience sample of patients seen at 2 medical centers. Subjects were restricted to those who could complete Quality of Life forms in Spanish or English.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No